CLINICAL TRIAL: NCT00395642
Title: TRIAGE-CRT Telemonitoring in Patients With Congestive Heart Failure and Indication of ICD-Cardiac Resynchronization Therapy
Brief Title: TRIAGE-CRT Telemonitoring in Patients With CHF and Indication of CRT-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Katerina de Metz / Director, Clinical Studies, Biotronik, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061653
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Congestive Heart Failure; Cardiac Resynchronization Therapy
Keywords: Congestive Heart Failure; Cardiac Resynchronization Therapy; Home Monitoring; Telemonitoring; Remote Monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM with weight and BP remote monitoring (Experimental): Device based Home Monitoring and weight and blood pressure remote monitoring
  Interventions: Device: Kronos LV-T, Lumax HF-T

INTERVENTIONS:
Device: Kronos LV-T, Lumax HF-T — Implanted CRT-device sends out device diagnostics (e.g. heart rate, device and lead integrity, patient activity) via CardioMessenger on daily basis. In addition, daily weight and blood pressure readings are taken; remote data are analyzed by investigational sites via the internet on a weekly basis.

SUMMARY:
This feasibility study will investigate the clinical benefit of the combined use of BIOTRONIK Home Monitoring (HM) and weight and blood pressure (BP) external telemonitoring (ETM) in the follow-up treatment of patients implanted with a Cardiac Resynchronization Therapy Implantable Cardioverter Defibrillator (CRT-D). The feasibility study is designed to plan and define endpoints for a larger randomized study. The study will assess the HM-parameter trends correlation with daily weight and blood pressure changes. The patient compliance rate of the two different telemonitoring systems (HM & ETM) will also be evaluated.

DETAILED DESCRIPTION:
This single-arm, multi-center feasibility study will explore the clinical benefit of the combined use of BIOTRONIK Home Monitoring (HM) and weight and blood pressure (BP) external telemonitoring (ETM) in the follow-up management of heart failure patients implanted with a Cardiac Resynchronization Therapy Implantable Cardioverter Defibrillator (CRT-D). The BIOTRONIK Home Monitoring system will automatically and remotely collect device based information on a daily basis, and an external telemonitoring system will be used to determine the 'weight' and 'blood pressure' remotely at the patient's home on a daily basis. This study will evaluate retrospectively, if Home Monitoring parameters correlate with weight and blood pressure changes. The patient compliance rate of the two telemonitoring systems will also be assessed.

Target enrollment is up to 100 patients at 15 U.S. sites. Patients will be enrolled within a period of 12 to 15 months. Based on the follow-up period of 6 months per patient, the study duration is 18 to 21 months from the date of first patient enrollment. All patients will give written informed consent prior to enrollment and will be implanted with the legally marketed BIOTRONIK Kronos LV-T, or an appropriate BIOTRONIK CRT-D, as well as legally marketed pacing and defibrillation leads. In addition, all patients will be receiving a legally marketed external telemonitoring system to determine weight and blood pressure at home.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Implanted within the past 45 days or being considered for implant with a BIOTRONIK CRT-D
* Age 18 years
* Able to follow and comply with the study related procedures
* Phone jack with landline connection at home to connect both the BIOTRONIK HM and the ETM system
* Sufficient cognitive and reading skills to operate weight & BP system Ambulatory
* Weight ≤ 400 lbs

Exclusion Criteria:

* Participation in another cardiovascular clinical study
* Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Akar, MD, Principal Investigator — Loyola University
Locations (12):
- United States (12):
  - Maricopa Medical Center, Phoenix, Arizona
  - Scottsdale Cardiology, Scottsdale, Arizona
  - Christiana Care Health Services, Wilmington, Delaware
  - Piedmont Hospital, Atlanta, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Loyola University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Thoracic & Cardiovascular Institute, Lansing, Michigan
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Cleveland Cardiovascular Research Foundation, Cleveland, Ohio
  - Pee Dee Cardiology, Florence, South Carolina
  - Spartanburg Regional, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Monitoring With Weight and BP Remote Monitoring: Device based Home Monitoring with weight and blood pressure (BP) remote monitoring
Period: Overall Study
Arm/Group | Home Monitoring With Weight and BP Remote Monitoring
Started | 66
Completed | 53
Not Completed | 13
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Home Monitoring With Weight and BP Remote Monitoring
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Patient Compliance of Weight and Blood Pressure External Monitoring and Home Monitoring Transmissions. Percentage of Days Transmitted.
Description: Analyzed transmission periods for weight, blood pressure (BP) and Home Monitoring (HM) started with the respective first transmission. In patients where neither system transmitted data, the date of enrollment was taken as the start date of the analyzed period for all systems. If only one remote system transmitted data (e.g. HM or weight and BP data only), the first transmission date from the corresponding, successfully transmitting system was assumed as the start date of the analyzed period for the non-transmitting system. Analyzed transmission period ended with study exit or completion.
Time Frame: 6 months
Population: All Enrolled Participants
Measure: Number; unit: Percent of days
Arm/Group | Home Monitoring With Weight and BP Remote Monitoring
Number analyzed (Participants) | 66
Percent of days
  Weight Telemonitoring | 71
  BP Telemonitoring | 71
  HM System | 83

ADVERSE EVENTS:
Arm/Group | Home Monitoring With Weight and BP Remote Monitoring
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 12/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Monitoring With Weight and BP Remote Monitoring (N=66)
Heart Failure related Hospitalization (Cardiac disorders) | 6 (9) — Adverse event with cardiac cause and resulted in or required treatment in hospital or an outatient setting (e.g. emergency room).
Death (General disorders) | 4 (4)
Complication (Cardiac disorders) | 3 (4) — Device related adverse event that required an invasive intervention to restore the function of the CRT-system (e.g. lead revision)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit copies of any proposed publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may delete any Confidential Information or other proprietary information. In addition, Sponsor may extend such review period for another 90 days to file patent applications or take other steps to protect its intellectual property interests.